CLINICAL TRIAL: NCT02452359
Title: Clinical Evaluation of Venus Versa SR Applicator Using Intense Pulsed Light on Skin Texture for Improving the Appearance of Striae Distensae
Brief Title: Clinical Evaluation of Using Intense Pulsed Light for Improving the Appearance of Striae Distensae
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Continuing the trial was considered to be superfluous.
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0315
Record Dates: First submitted 2015-05-08; First posted 2015-05-22 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Striae Distensae
Keywords: stretch marks
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Intervention Model Description: Open-label study where all subjects assigned to receive 5 treatments every 2 weeks. Subjects acted as their own control.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Group (Experimental): Group receiving treatment with Venus Versa IPL energy
  Interventions: Device: Venus Versa

INTERVENTIONS:
Device: Venus Versa — The Venus Versa system consists of a console and 4 detachable applicators that deliver optical energy in the form of Intense Pulsed Light to the patient skin. The intense pulsed light lamp delivers non-coherent light distributed over a range of wavelengths from 500 nm to 1200 nm. Different filters are embedded in the different applicators so that each applicator can deliver the desired spectrum according to the indications to be treated.In this study, the IPL applicator SR580 will be evaluated for the treatment of Striae Distensae, depending on the patient's skin type.

SUMMARY:
This trial is intended to evaluate the effect of IPL treatment on the Striae Distensae. The study hypothesis is that the SR580 applicator will improve the appearance of Striae Distensae by at least 1 point on the Global Aesthetic Improvement ScaleI (GAIS) at 3 months follow-up compared to baseline in at least 50% of the study population.

DETAILED DESCRIPTION:
Study Design This is a multi-site, prospective, open labeled clinical trial with before-after study design. This study will include up to 8 visits at the clinic: initial screening/consultation, 5 treatments, visits in 2 week intervals, and 2 follow-up visits at 1 and 3 months after the last treatment visit.

Up to 60 healthy subjects age 24-65 with Striae Distensae will be enrolled.

Study duration:

Duration of subject's participation: Up to 5.5 months from enrollment to termination

Blinding Objective assessment of clinical improvement by global assessment scale will be achieved by sending before/after pictures (baseline/3months after last treatment) to 3 blinded reviewers at the end of the study.

Study Procedures Test Spots Up to 3 test spots will be performed in the selected treatment area to determine the optimal parameters / settings

Treatment visits Each subject will be enrolled and scheduled for 5 treatments at 2 week intervals and return for follow-up visits at one month and 3 months after the last treatment for evaluation of the treated areas. The duration of the entire treatment visit is approximately 60 minutes.

Treatment The treatment areas are divided into 2 treatment areas: abdomen or thighs. Apply a thin layer of IPL gel. Place the applicator in close contact, perpendicular to the skin with no pressure applied. Pressing the applicator will fire the IPL pulse.

Administer pulses throughout the treated area to ensure full coverage of the treated area with applicator overlap approximately 1/3 of the previously treated skin.

A single pass over the area is completed Remove the remnants of the IPL gel and dry thoroughly. Cold air or cold, wet but not frozen gauze pads may be placed on the treated area for post treatment cooling.

Typical responses to the treatment are mild erythema and edema.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written Informed Consent;
2. Healthy male or female, 24-65 years Fitzpatrick-Goldman skin type I-V;
3. Having visible Striae Distensae to be treated (abdomen/thighs);
4. Comply with the treatment/follow-up schedule and requirements;
5. Women of child-bearing age are required to be using a reliable method of birth control

Exclusion Criteria:

1. Fitzpatrick-Goldman skin type VI;
2. Pregnant, intending to become pregnant during the course of study, less than 3 months postpartum or less than 6 weeks after breastfeeding;
3. Heavy smoker
4. Unable or unlikely to refrain from tanning
5. Use of photosensitive medication
6. Use of oral isotretinoin within 3 months
7. Any dermal/epidermal damage or disorder in treated area
8. Prior treatment in treated area within 3 months
9. Prior skin laser/light or another device treatment in treated area within 6 months
10. Prior use of collagen, fat injections or other methods of skin augmentation in treated area within 12 months
11. Prior use of Botox in treatment area within 6 months
12. Prior ablative resurfacing procedure with laser in treatment area within 12 months
13. Any other surgery in treated area within 9 months
14. Participation in a study of another investigational device or drug as per the Investigator's discretion
15. History of keloid or any other type of hypertrophic scar formation or poor wound healing in a previously injured skin area
16. Showing symptoms of hormonal disorders (such as Melasma, Chloasma);
17. Concurrent inflammatory skin conditions, open laceration or abrasion of any sort on area to be treated during the course of treatment
18. Active Herpes Simplex at the time of treatment or having experienced more than three episodes of Herpes Simplex eruption within a year of study
19. Multiple dysplastic nevi in area to be treated
20. Having a bleeding disorder or taking anticoagulation medications
21. History of immunosuppression/immune deficiency disorders
22. Having any form of active cancer at the time of enrollment and during the course of the study or history of skin cancer
23. Pigmented lesion in the treated area that appears cancerous
24. Significant concurrent illness, such as uncontrolled diabetes
25. Active infections in the treated area

28.Tattoo or permanent makeup at the treatment area. 29.Mentally incompetent, prisoner or evidence of active substance or alcohol abuse 30.Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-03-13 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey L Mancuso, Study Director — Venus Concept
Locations (1):
- Rosenberg Plastic Surgery, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each subject to receive IPL 580 nm treatment to striae distensae on either abdomen or thighs. Baseline photos taken of untreated treatment area.
Groups:
- IPL 580 nm Treatment: Each subject to receive IPL applicator SR580 treatment of Striae Distensae either on the abdomen or thighs.
Period: Overall Study
Arm/Group | IPL 580 nm Treatment
Started | 54
Completed | 33
Not Completed | 21
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 15
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Group receiving treatment with Venus Versa IPL energy
  Venus Versa: The Venus Versa system consists of a console and 4 detachable applicators that deliver optical energy in the form of Intense Pulsed Light to the patient skin. The intense pulsed light lamp delivers non-coherent light distributed over a range of wavelengths from 500 nm to 1200 nm. Different filters are embedded in the different applicators so that each applicator can deliver the desired spectrum according to the indications to be treated.In this study, the IPL applicator SR580 will be evaluated for the treatment of Striae Distensae, depending on the patient's skin type.
  IPL gel: water based gel used to protect the skin during light based treatments. Is also commonly used during ultrasound treatments.
Arm/Group | Treatment Group
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1
  Female | 32
  Unknown | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 6
  Caucasian | 25
  Other | 1
  unknown | 22
Baseline photograph of treatment area [Count of Participants; unit: Participants] — Body area with visible Striae Distensae, either abdomen or thighs. Population: The baseline photographs were not evaluated.

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Striae Distensae Appearance
Description: Striae distensae appearance improvement by at least 1 point on the Global Aesthetic Improvement scale (GAIS) from photographs 3 months following the last treatment as determined by 3 blinded reviewers where 3 = Very Much Improved, 2 = Much Improved, 1 = Improved, 0 = No Change, -1 = Worse, -2 = Much Worse and -3 = Very Much Worse.
Time Frame: 90 days following last IPL treatment
Population: The primary outcome measure is not reported as data not collected.
Groups:
- Treatment Group: Group receiving treatment with Venus Versa IPL energy
  Venus Versa: The Venus Versa system consists of a console and 4 detachable applicators that deliver optical energy in the form of Intense Pulsed Light to the patient skin. The intense pulsed light lamp delivers non-coherent light distributed over a range of wavelengths from 500 nm to 1200 nm. Different filters are embedded in the different applicators so that each applicator can deliver the desired spectrum according to the indications to be treated.In this study, the IPL applicator SR580 will be evaluated for the treatment of Striae Distensae, depending on the patient's skin type.
  IPL gel: water based gel used to protect the skin during light based treatments.
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year 11 months
Groups:
- IPL 580 nm Treatment: All subjects who received at least one IPL treatment.
Arm/Group | IPL 580 nm Treatment
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT02452359/Prot_SAP_000.pdf